CLINICAL TRIAL: NCT05097521
Title: Complementary and Integrative Health for Pain in the VA: A National Demonstration Project (NIH-VA-DOD Joint Initiative)
Brief Title: Assessing Pain, Patient Reported Outcomes and Complementary and Integrative Health
Acronym: APPROACH
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Veterans Health Administration Office of Patient Centered Care & Cultural Transformation (Unknown)
Responsible Party: Sponsor
Other Study IDs: SDR 17-306
Record Dates: First submitted 2021-10-14; First posted 2021-10-28 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Complementary Therapies; Chronic Pain; Integrative Medicine; Chiropractic; Acupuncture; Yoga; Tai Chi; Meditation
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy; Massage; Yoga; Meditation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Veterans using practitioner delivered CIH therapies only: Veterans using practitioner-delivered (acupuncture, chiropractic care, massage) CIH therapies only
  Interventions: Other: Practitioner-delivered CIH therapies (acupuncture, therapeutic massage, chiropractic care) as received in VHA and community practice settings
- Veterans using self-care CIH therapies only: Veterans using self-care (yoga, meditation, Tai Chi, Qi Gong) CIH therapies only
  Interventions: Other: Self-care CIH therapies (yoga, Tai Chi/Qigong , meditation) as received in VHA and community practice settings
- Veterans using a combination of practitioner-delivered and self-care CIH therapies (dual-care): Veterans using a combination of practitioner-delivered and self-care CIH therapies (dual-care)
  Interventions: Other: Combination of practitioner-delivered and self-care CIH therapies (described above) as received in VHA and community practice settings

INTERVENTIONS:
Other: Practitioner-delivered CIH therapies (acupuncture, therapeutic massage, chiropractic care) as received in VHA and community practice settings — Practitioner-delivered CIH therapies (acupuncture, therapeutic massage, chiropractic care) as received in VHA and community practice settings
  Groups: Veterans using practitioner delivered CIH therapies only
Other: Self-care CIH therapies (yoga, Tai Chi/Qigong , meditation) as received in VHA and community practice settings — Self-care CIH therapies (yoga, Tai Chi/Qigong , meditation) as received in VHA and community practice settings
  Groups: Veterans using self-care CIH therapies only
Other: Combination of practitioner-delivered and self-care CIH therapies (described above) as received in VHA and community practice settings — Combination of practitioner-delivered and self-care CIH therapies (described above) as received in VHA and community practice settings
  Groups: Veterans using a combination of practitioner-delivered and self-care CIH therapies (dual-care)

SUMMARY:
The APPROACH Study (Assessing Pain, Patient-Reported Outcomes and Complementary and Integrative Health) assesses the effects of use of practitioner-delivered CIH therapies alone compared to the combination of self-care and practitioner-delivered CIH therapies among Veterans with chronic musculoskeletal pain. The APPROACH study is predominately conducting a secondary analysis of patient-reported data being collected by the Veterans Health Administration's (VA) Office of Patient Centered Care and Cultural Transformation among Veterans using 18 VA medical centers. Those facilities received funding as part of the Comprehensive Addiction and Recovery Act to expand availability of CIH therapies. That patient-reported data is being supplemented with VA electronic health record data and data on the 18 medical centers' business practices (nudges, the instrumental variable). Practitioner-delivered therapies under study include chiropractic care, acupuncture and therapeutic massage, and self-care therapies include Tai Chi/qigong, yoga and meditation. The primary outcomes are improvement in pain severity and pain interference, using the Brief Pain Inventory (BPI), 6 months after initiating CIH therapies compared to baseline. Patients will enter treatment groups based on the CIH therapies they use, as randomizing patients to specific therapies would require withholding therapies routinely offered at VA. The investigators will address selection bias and confounding by using sites' variations in business practices and other encouragements (nudges) to receiving different CIH therapies as a surrogate for direct randomization using instrumental variables econometric methods.

DETAILED DESCRIPTION:
Design: The investigators are employing a quasi-experimental encouragement study design in which subjects are able to choose their own CIH therapies, but some are offered extra encouragements (nudges) to choose specific CIH therapies. Instead of being randomized to a CIH therapy, individuals will enter one of the two study groups based on what CIH therapies they used six months after they initiate any CIH therapy. Although accrual to study group is not random, some sites have strong business practices/nudges that lead to considerable variation in which CIH therapies patients use. The variation induced by these business practices/nudges provides a quasi-experimental natural experiment that can be assessed through an instrumental variables analytic approach. The purpose of using business practices as an instrument for accruing patients to treatment group, similar to the use of randomization, is to reduce potential selection and confounding bias. The 6-month treatment window will allow for patients to initiate one type of CIH therapy and add additional CIH therapies based on business practices/nudges at their site within the evaluation period. The CIH therapies that patients receive will be as they are delivered by the 18 VHA Whole Health flagship study sites and community care practices.

Sites: The study sites are the VA's 18 Whole Health Flagship sites: VA Boston Health Care System, VA New Jersey Health Care System, Erie VAMC, Beckley VAMC, W. G. (Bill) Hefner VAMC, Atlanta VAMC, Tampa VAMC, Tennessee Valley Health Care System, Aleda E. Lutz VAMC, Tomah VAMC, St. Louis VA Health Care System, Central Arkansas Veterans Healthcare System, South Texas Veterans Health Care System, Salt Lake City VAMC, VA Portland Health Care System, Palo Alto VAMC, Tucson VAMC, VA Nebraska-Western Iowa Health Care System).

Secondary Data from the CIH Experience Survey/ VA Office of Patient Centered Care and Cultural Transformation's Survey: The APPROACH study is predominately conducting a secondary analysis of patient-reported data being collected by VA OPCC&CT's survey. That is a 4-time point survey (baseline and months 1, 3, 6). Almost all of the outcomes listed below are from that survey.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* History of (chronic) musculoskeletal-related pain conditions recorded in the EHR in the year prior to the index visit, and self-report pain present every day or nearly every day for 3 months from the CIH index visit using an eligibility screener
* 18-89 on index CIH visit date

Exclusion Criteria:

* diagnoses of serious mental illness in the year prior to initiating CIH
* history of spinal cord injury
* hospitalization 30 days prior to initiating CIH
* recorded CIH use in the EHR in the 6 months prior to the index CIH visit and reported CIH use in the 8 weeks prior to index CIH visit

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe chronic musculoskeletal pain who initiate at least one of the six CIH therapies at the 18 VA Whole Health flagship study sites during the study period who also participate in the VA Office of Patient Centered Care and Cultural Transformations CIH Experience Survey.
Sampling Method: Non-Probability Sample
Enrollment: 3726 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-09-17 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory Interference Scale | Change from baseline to 6 months
  Measure of pain-related functional interference. Scores range 0-10; higher score is worse.
Brief Pain Inventory Severity Scale | Change from baseline to 6 months
  Measure of pain intensity. Scores range 0-10; higher score is worse.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) for improvement in pain | baseline, 1 month, 3 months, and 6 months
  Scores range 1-5; 1=much better, 5 = much worse.
Patient Global Impression of Change (PGIC) for improvement in mental health | 6 months
  Scores range 1-5; 1=much better, 5 = much worse.
Patient Global Impression of Change (PGIC) for improvement in physical health | 6 months
  Scores range 1-5; 1=much better, 5 = much worse.
Patient Global Impression of Change (PGIC) for improvement in fatigue | 6 months
  Scores range 1-5; 1=much better, 5 = much worse.
Patient Global Impression of Change (PGIC) for improvement in overall well-being | 6 months
  Scores range 1-5; 1=much better, 5 = much worse.
PROMIS10 global assessment of physical health | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating better health.
PROMIS10 global assessment of mental health | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating better health.
PROMIS10 assessment of fatigue | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating better health.
PROMIS10 assessment of general quality of life | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating better health.
Life Engagement Test (LET) | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating better life engagement.
Perceived Stress Scale (PSS-4) | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating more perceived stress.
Patient Health Questionnaire (PHQ2) | Change from baseline to 6 months
  Measure of depressed mood and anhedonia. Scores range from 0 to 6, with higher scores indicating more depressive symptoms.

OTHER OUTCOMES:
Perceived Health Competency Scale (PHCS-2) | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating lower perceived health competency.
Altarum Consumer Engagement (ACE) | Change from baseline to 6 months
  Items are rated on a five-point scale with higher scores indicating lower patient engagement.
Self-Efficacy for Managing Chronic Disease (SEMCD) | Change from baseline to 6 months
  Items are rated on a ten-point scale with higher scores indicating higher self-efficacy. Only items 5 and 6 are included in the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Taylor, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA; Steven B. Zeliadt, PhD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
The APPROACH study is primarily a study of existing data. As such, the investigators will not have data to share.

REFERENCES:
- [Background] Zeliadt SB, Coggeshall S, Thomas E, Gelman H, Taylor SL. The APPROACH trial: Assessing pain, patient-reported outcomes, and complementary and integrative health. Clin Trials. 2020 Aug;17(4):351-359. doi: 10.1177/1740774520928399. Epub 2020 Jun 10. PMID 32522024
- [Background] Zeliadt SB, Coggeshall S, Gelman H, Shin MH, Elwy AR, Bokhour BG, Taylor SL. Assessing the Relative Effectiveness of Combining Self-Care with Practitioner-Delivered Complementary and Integrative Health Therapies to Improve Pain in a Pragmatic Trial. Pain Med. 2020 Dec 12;21(Suppl 2):S100-S109. doi: 10.1093/pm/pnaa349. PMID 33313736
- [Background] Ali J, Antonelli M, Bastian L, Becker W, Brandt CA, Burgess DJ, Burns A, Cohen SP, Davis AF, Dearth CL, Dziura J, Edwards R, Erdos J, Farrokhi S, Fritz J, Geda M, George SZ, Goertz C, Goodie J, Hastings SN, Heapy A, Ilfeld BM, Katsovich L, Kerns RD, Kyriakides TC, Lee A, Long CR, Luther SL, Martino S, Matheny ME, McGeary D, Midboe A, Pasquina P, Peduzzi P, Raffanello M, Rhon D, Rosen M, Esposito ER, Scarton D, Hastings SN, Seal K, Silliker N, Taylor S, Taylor SL, Tsui M, Wright FS, Zeliadt S. Optimizing the Impact of Pragmatic Clinical Trials for Veteran and Military Populations: Lessons From the Pain Management Collaboratory. Mil Med. 2022 Jul 1;187(7-8):179-185. doi: 10.1093/milmed/usab458. PMID 34791412
- [Background] Der-Martirosian C, Shin M, Upham ML, Douglas JH, Zeliadt SB, Taylor SL. Telehealth Complementary and Integrative Health Therapies During COVID-19 at the U.S. Department of Veterans Affairs. Telemed J E Health. 2023 Apr;29(4):576-583. doi: 10.1089/tmj.2022.0209. Epub 2022 Jul 22. PMID 35867052
- [Background] Kerns RD, Davis AF, Fritz JM, Keefe FJ, Peduzzi P, Rhon DI, Taylor SL, Vining R, Yu Q, Zeliadt SB, George SZ. Intervention Fidelity in Pain Pragmatic Trials for Nonpharmacologic Pain Management: Nuanced Considerations for Determining PRECIS-2 Flexibility in Delivery and Adherence. J Pain. 2023 Apr;24(4):568-574. doi: 10.1016/j.jpain.2022.12.008. Epub 2022 Dec 24. PMID 36574858